CLINICAL TRIAL: NCT04367376
Title: The Short-term Effects of Instrument-Based Mobilization Compared With Manual Mobilization for Low Back Pain: A Randomized ClinicalTrial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Fadela Alqassab, Ms., Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-PGS-2018-03-286
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain, Mechanical
MeSH Terms: conditions — Low Back Pain | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- manual therapy (Experimental): The control group will receive central postero-anterior grade III mobilization through the pisiform grip method at the level of pain in the lumbar spine.
  Interventions: Other: mobilization; Other: manual therapy
- instrumental manual therapy (Experimental): the intervention groub rcieved central postero-anterior mobilization with a force of 20-30 N through physiotherapy instrument mobilization at the level of pain in the lumbar spine.
  Interventions: Other: mobilization; Other: instrumental manual therapy

INTERVENTIONS:
Other: mobilization — central postroanterion mobilization on the most painful vertebral level at the lumbar spine
Other: manual therapy — manual therapy
  Arms: manual therapy
Other: instrumental manual therapy — instrumental manual therapy
  Arms: instrumental manual therapy

SUMMARY:
Objectives: To investigate the effectiveness of instrument-based mobilization compared with manual mobilization in patients with non-specific low back pain (NLBP), in terms of spinal muscle activation, decrease in pain, and improvement in range of motion (ROM).

Design: Randomized clinical trial, double blind. Participants and interventions: A total of 66 participants with localized NLBP will be divided into 2 groups matched for sex, age, and body mass index. The intervention group will receive central postero-anterior mobilization with a force of 150 N through physiotherapy instrument mobilization at the level of pain in the lumbar spine. The control group will receive central postero-anterior grade III mobilization through the pisiform grip method at the level of pain in the lumbar spine.

Main outcome measures: Measurements will be taken before the intervention, after the 1st session, after the 6th session, and at 4 weeks follow-up. Rehabilitative ultrasound imaging will be done to identify lumbar multifidus (LM) activation through the measurement of muscle thickness at the level of L5-L4 vertebrae, during rest and lower-extremity movement. Each participant will self-rate the pain intensity in the lumbar spine according to the Numeric Pain Rating Scale (NPRS). The pressure-pain threshold (PPT) will be measured using an algometer. Lumbar ROM will be measured using a dual inclinometer method in flexion and extension.

The results will be compared between the intervention and control groups through mixed analysis of variance for LM thickness, lumbar ROM, PPT, and NPRS.

ELIGIBILITY:
Inclusion Criteria:

* age 20-59 years (commonly affected age range), BMI 18.5-30 kg/m2 (normal to overweight), localized NLBP, pain duration <12 months, and pain score ≥3/10 on the NPRS.

Exclusion Criteria:

* history of spinal surgery, significant previous back trauma, spinal or lower-extremity deformities, LBP associated with peripheral neurological symptoms (paraesthesia, anaesthesia, signs of nerve root compression), neurological diseases, systemic diseases (diabetes mellitus, rheumatoid arthritis), and any contraindication to manual therapy (spinal instability, healing fracture, dislocations, pregnancy in women).

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 2-3 weeks
  a series of numbers from 0 to 10, with '0' indicating no pain and '10' indicating the most intense pain possible
Lumbar Multifidus muscle activation | 2-3 weeks
  muscle activation quantified by measuring the muscle thickness during rest and activation positions.

SECONDARY OUTCOMES:
Pressure pain threshold | 2-3 weeks
  measured at the most painful site on the back as well as on a mid-point at RT tibialis anterior muscle belly lateral to the tibia
Lumbar spine ROM | 2-3 weeks
  measured in flexion, extension, and lateral flexion to both sides. Dual inclinometer method used to take the measurements (Baseline Bubble Inclinometer device)

CONTACTS AND LOCATIONS:
Locations (1):
- Imam Abdulrahman Bin Faisal University, Khobar, Eastern Province, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No